CLINICAL TRIAL: NCT00297141
Title: Preoperative Combined Radiochemotherapy for Patients With Newly Diagnosed, Primary Operable and Locally Advanced Rectal Carcinoma (cT3, Nx, M0) of the Lower and Middle Rectum
Brief Title: Preoperative Combined Radiochemotherapy for Patients With Rectal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Collaborators: Sanofi-Synthelabo (Industry); Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABCSG 95 / TAKO 05; Studie R02 (95) (Other: ABCSG internal study code); 2004-002358-72 (EudraCT Number)
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Rectal Cancer
Keywords: Preoperative; Radiochemotherapy; Newly Diagnosed; Primary Operable; Locally Advanced; Rectal Carcinoma; T3; Lower Rectum; Middle Rectum; ABCSG; TAKO; 95; 05
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm (radiochemotherapy) (Experimental): single arm study (capecitabine, oxaliplatin)
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Capecitabine — chemotherapy oral use
  Other Names: Xeloda; RO 09-1978
Drug: Oxaliplatin — chemotherapy intravenous use
  Other Names: treatment defined only by active substance; (no trade name defined; investigators choice)

SUMMARY:
Rate of T-downstaging (Reduction of the T-stadium) at the time of final surgery following the preoperative combined radiochemotherapy (chemotherapy: Oxaliplatin, Capecitabine) Evaluation of the toxicity grade III and IV of the therapy scheme

DETAILED DESCRIPTION:
About 60 patients with locally advanced rectal carcinoma (cT3, Nx, M0) of the lower and middle rectum will be recruited.

The radiotherapy is an essential part of therapy of the advanced rectal carcinoma and the additional administration of a chemotherapy will positively influence the effect of the therapy (downstaging-rate, rate of distant metastases, survival-rate). Probably a downsizing and downstaging (as per literature and by own experience) can be reached with an preoperative combined radiochemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 80
* Biooptical confirmed adenocarcinoma of the lower und middle rectum (lower edge of the tumor located max. 14 cm of the anal verge)
* According to MRI tumor extensions into the perirectal fat tissue (cT3)
* No former chemotherapy, radiotherapy and/or tumor resection of a rectum carcinoma
* WHO performance status 0 - 2
* Adequate bone marrow reserve (leucocytes - not more than 3.000/ml; thrombocytes - not more than 100.000/ml)
* Adequate hepatic function (bilirubin - not more than 1.5 x ULN; GOT and GPT - not more than 3.5 x ULN)
* Adequate renal function (creatinin - not more than 1.5 mg/dl)
* Women of childbearing potential: exclusion of pregnancy (negative urin or serum pregnancy test)
* Willingness of women of childbearing potential and accordingly of potent men to use approved contraceptives (for example birth-control pill, loop, condom) during and at least 3 month after closure of the study
* Life expectancy of at least 3 month
* Signed written Informed Consent before recruitment
* Exclusion of distant metastases at the time of recruitment

Exclusion Criteria:

* Former radio- and/or chemotherapy
* Tumor of the upper rectum
* Any other kind of malign tumor in the last five years (except adequate treated basal cell carcinoma of the skin, or in situ cervical carcinoma)
* Peripheral Neuropathy (NCI CTC - not higher than Grade 1)
* General contraindication or hypersensitivity against Oxaliplatin and/or Capecitabine
* Any other untreated not malign diseases: Cardiac insufficiency, angina pectoris, hypertension or arrhythmia, hepatic diseases, significant neurological or psychiatric disorders
* Florid, serious infection at the time of recruitment
* Legally limited capacity or evidence of a neurological or psychiatric disease, the investigator is the opinion it will constrict the patients compliance
* Evidence of lacking willingness for cooperation of the patient
* Pregnant or breast feeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2004-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Rate of T-downstaging (Reduction of the T-stadium) | at the time of final surgery
  surgery following the preoperative combined radiochemotherapy (chemotherapy: Oxaliplatin, Capecitabine)

SECONDARY OUTCOMES:
Evaluation of the toxicity grade III and IV of the therapy scheme | week 1 to max. week 10
  from Visit 1 till surgery: weekly visits (visit 1 to visit 5) followed by final examination (performed 1 to 2 weeks after visit 5) before surgery followed by hospital admission (performed 1 to 2 weeks after final examination) followed by surgery ((performed 1 to 2 weeks after hospital admission)

CONTACTS AND LOCATIONS:
Overall Officials: Dietmar Oefner, MD, Principal Investigator — Austrian Breast & Colorectal Cancer Study Group; Alexander de Vries, MD, Principal Investigator — Austrian Breast & Colorectal Cancer Study Group; Josef Thaler, MD, Principal Investigator — Austrian Breast & Colorectal Cancer Study Group
Locations (8):
- Austria (8):
  - Hospital BHB St. Veit/Glan, Surgery, Saint Veit A. D. Glan, Carinthia
  - Hospital Wiener Neustadt, Wiener Neustadt, Lower Austria
  - Paracelsus Medical University Salzburg - Oncology, Salzburg, Salzburg
  - Medical University of Graz, Oncology, Graz, Styria
  - State Hospital Leoben, Surgery, Leoben, Styria
  - Medical University of Innsbruck, Surgery, Innsbruck, Tyrol
  - Klinikum Wels-Grieskirchen GmbH, Wels, Upper Austria
  - Medical University of Vienna, Radiotherapy, Vienna, Vienna

REFERENCES:
- [Derived] Ofner D, Devries AF, Schaberl-Moser R, Greil R, Rabl H, Tschmelitsch J, Zitt M, Kapp KS, Fastner G, Keil F, Eisterer W, Jager R, Offner F, Gnant M, Thaler J; TAKO 05/ABCSG R-02 Trial Investigators. Preoperative oxaliplatin, capecitabine, and external beam radiotherapy in patients with newly diagnosed, primary operable, cT(3)NxM0, low rectal cancer: a phase II study. Strahlenther Onkol. 2011 Feb;187(2):100-7. doi: 10.1007/s00066-010-2182-6. Epub 2011 Jan 21. PMID 21267531